CLINICAL TRIAL: NCT02458131
Title: TEEN HEED: An Adolescent Peer Led Diabetes Prevention Intervention
Brief Title: Community-based Adolescent Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GCO 13-0901; 5K23DK101692-02 (NIH)
Record Dates: First submitted 2015-05-22; First posted 2015-05-29 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Pre-Diabetes
Keywords: community-based participatory research; adolescents
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEEN HEED (Experimental): Adolescent pre-diabetics will receive 8-12 weekly peer-led diabetes prevention educational workshops in community sites. The in-person group workshops will be supplemented by support through mobile health technologies such as text messaging and social media.
  Interventions: Behavioral: TEEN HEED
- Wait List Control (No Intervention): Adolescent pre-diabetics in this group will not receive any intervention until collection of all follow up data and will then be offered the same intervention as the participants in the experimental arm.

INTERVENTIONS:
Behavioral: TEEN HEED — Peer-led workshops will cover behavioral skills including goal setting, self-monitoring, problem solving, contingency management, coping skills, and social support.
  Arms: TEEN HEED

SUMMARY:
The number of youth with type 2 diabetes is predicted to quadruple by 2050, with a disproportionate increase among minority youth. The research proposed in this Career Development Award will use community-based participatory research methodology as well as novel strategies (peer education and mobile health technologies) to design, implement and evaluate a diabetes prevention intervention for at-risk ethnic minority youth in an urban community with high disease burden.

DETAILED DESCRIPTION:
Approach: The proposed research addresses diabetes risk and prevention among racial/ethnic minority adolescents in East Harlem (EH), NY. Aim 1 will use qualitative methods to explore the best strategies for using peer education for diabetes risk reduction in youth and the potential role of mobile health technologies in improving adherence to behavioral modification plans. Aim 2 will utilize findings from preliminary studies and Aim 1 to design and evaluate a pilot community-based intervention to 1) maintain/reduce BMI (primary outcome), 2) improve adolescent dietary, physical activity and weight control behaviors, and 3) improve other measures of diabetes risk. Data will be collected at baseline, immediately after the intervention (3 months) and at one year in the intervention and wait list control groups. Aim 3 involves refining the pilot intervention based on an examination of intervention feasibility, acceptability, and sustainability and planning for a future R01.

ELIGIBILITY:
Inclusion Criteria for pre-diabetes screening:

* Adolescents ages 13-19 years of age
* English speaking
* Residents of East Harlem or members of an East Harlem Institution. Membership in an East Harlem institution includes the following:

  1. attending a school in East Harlem
  2. attending an after school or recreational activity in East Harlem
  3. receiving health care in East Harlem Proof of address or membership in an East Harlem institution will not be asked.
* At risk for diabetes (overweight/obese based on measured BMI percentile and with either a parent or grandparent with type 2 diabetes)
* No plans to relocate from New York City in the next year

Note: additional inclusion criteria for participation in workshops include diagnosis of pre-diabetes based on oral glucose tolerance test

Exclusion Criteria for pre-diabetes screening:

* <13 or >19 years of age
* Previous diagnosis of diabetes
* BMI percentile <85th percentile for age and gender based on Centers for Disease Control and Prevention definition
* Currently pregnant
* Speaking a language other than English
* On medications that may raise or lower blood sugar
* Plans to relocate from New York City within one year of enrollment-

Note: additional exclusion criteria for participation in workshops include fingerstick glucoses outside the pre-diabetes range during oral glucose tolerance testing and any cognitive or physical impairment that would preclude comprehension of the group educational program

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2019-08-24 (Actual); Study Completion 2019-08-24 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | Baseline and 3 months
  Change in BMI at post-intervention (approximately 3 months) as compared to baseline
Change in BMI | Baseline and 1 year
  Change in BMI at 1 year as compared to baseline

SECONDARY OUTCOMES:
Change in fasting blood glucose levels | Baseline and 3 months
  Change in fasting blood glucose levels at post-intervention (approximately 3 months) as compared to baseline
Change in fasting blood glucose levels | Baseline and 1 year
  Change in fasting blood glucose levels at 1 year as compared to baseline
Change in post prandial blood glucose level | Baseline and 3 months
  Change in post prandial blood glucose level at post-intervention (approximately 3 months) as compared to baseline
Change in post prandial blood glucose level | Baseline and 1 year
  Change in post prandial blood glucose level at 1 year as compared to baseline
Change in blood pressure | Baseline and 3 months
  Change in blood pressure at post-intervention (approximately 3 months) as compared to baseline
Change in blood pressure | Baseline and 1 year
  Change in blood pressure at 1 year as compared to baseline
Change in percent body fat | Baseline and 3 months
  Change in percent body fat at post-intervention (approximately 3 months) as compared to baseline
Change in percent body fat | Baseline and 1 year
  Change in percent body fat at 1 year as compared to baseline
Change in waist circumference | Baseline and 3 months
  Change in waist circumference at post-intervention (approximately 3 months) as compared to baseline
Change in waist circumference | Baseline and 1 year
  Change in waist circumference at 1 year as compared to baseline
Change in knowledge, attitudes, beliefs and behaviors related to diabetes and weight loss | Baseline and 3 months
  Change in knowledge, attitudes, beliefs and behaviors (from the TEEN HEED survey) at post-intervention (approximately 3 months) as compared to baseline
Change in knowledge, attitudes, beliefs and behaviors related to diabetes and weight loss | Baseline and 1 year
  Change in knowledge, attitudes, beliefs and behaviors (from the TEEN HEED survey) at 1 year as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nita Vangeepuram, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States